CLINICAL TRIAL: NCT00487305
Title: A Phase I Trial of Vaccination With Lethally Irradiated Lymphoma Cells Admixed With Granulocyte-Macrophage Colony Stimulating Factor Secreting K562 Cells for the Treatment of Previously Untreated or Relapses Follicular Lymphoma
Brief Title: Vaccination for the Treatment of Previously Untreated or Relapsed Follicular Lymphoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Responsible Party: Principal Investigator, Eric Jacobsen, MD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 06-275
Record Dates: First submitted 2007-06-15; First posted 2007-06-18 (Estimated); Last update posted 2024-08-15 (Actual); Status verified 2024-08

CONDITIONS: Follicular Lymphoma
Keywords: GM-CSF; vaccine; K562
MeSH Terms: conditions — Lymphoma, Follicular

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Biological/Vaccine (Experimental): Biological/Vaccine: Lethally Irradiated Lymphoma cells with GM-CSF K562 Cells Dose will vary depending upon number of cells collected and when the participant is enrolled on the study: the vaccine is given as an injection under the skin once weekly for 3 weeks then every other week for 3 vaccines.
  --------------------------------------------------------------------------------
  Interventions: Biological: Lethally Irradiated Lymphoma cells with GM-CSF K562 Cells

INTERVENTIONS:
Biological: Lethally Irradiated Lymphoma cells with GM-CSF K562 Cells — Dose will vary depending upon number of cells collected and when the participant is enrolled on the study: the vaccine is given as an injection under the skin once weekly for 3 weeks then every other week for 3 vaccines.

SUMMARY:
The purpose of this study is to compare the safety and immune activity of three doses of tumor vaccine. In recent years, researchers at the Dana-Farber Cancer Institute have discovered that vaccines made from patient's own cancer cell, that have been engineered in the laboratory to produce a protein called GM-CSF, can be effective in stimulating a powerful immune response specific to that cancer. GM-CSF is a naturally occuring hormone in the body that helps our immune system fight infections and diseases. One of the goals of this study is to determine whether these vaccinations will improve the immune system's ability to recognize and destroy the participant's lymphoma cells.

DETAILED DESCRIPTION:
* The dose of vaccine will depend upon how many of the participant's own tumor cells are available and at which point they join study. This Phase I trial is a "dose escalation" study. This means that participants will be enrolled in groups. Group 2 will receive a larger dose than Group 1. Group 3 will receive a larger dose than Group 2.
* The vaccine is administered in injections under and into the skin six times. Participants will receive vaccination shots once weekly for 3 vaccines, then every other week for 3 vaccines.
* After the first and fifth vaccinations, a small amount of the participants own lymphoma cells (killed) will be injected under the skin to see if their immune system will react against it and cause redness and swelling. A punch skin biopsy will also be performed at these injection locations.
* During the course of the study, we will also be drawing blood to evaluate immune cells and the effect that the vaccinations have on the participants immune system. During all treatment cycles a physical exam and questions about the participants general health will be performed.
* After the final treatment (approximately week 10) the participant will undergo "re-staging" to assess the status of their disease. If after completion of six vaccines, evaluation of the participant's disease reveals that it is stable or responding to the vaccine, and there is still vaccine available, they may be eligible to continue to receive the vaccines every two weeks until their supply runs out.
* After completion of the vaccinations, participants will come back for physical exams and blood tests every 3 months for 1 year and then once a year for fifteen years to monitor the effects of the vaccine.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed follicular lymphoma
* Patients with relapsed follicular lymphoma achieving at least a PR following their most recent systemic chemotherapy and/or immunotherapy regimen.
* Lymphoma accessible for sampling or existing cryopreserved lymphoma tumor judged suitable for vaccine preparation.
* 4 weeks must have elapsed between the completion of the the last chemotherapy, immunotherapy, glucocorticoid therapy, radiotherapy, or experimental therapy.
* ECOG Performance Status 0 or 1
* Estimated life expectancy of > 6 months
* 35 years of age or older
* Adequate recovery of drug related toxicities, surgery or radiation therapy
* Greater than 6 months since autologous stem cell transplantation
* Laboratory parameters as outlined in the protocol

Exclusion Criteria:

* Uncontrolled active infection or illness
* Psychiatric illness/social situation that would limit study compliance
* Pregnancy or nursing mothers
* Evidence of infection with HIV or viral hepatitis
* Other invasive malignancy
* Existing autoimmune cytopenia
* Previous allogeneic stem cell transplant
* Pre-existing autoimmune disease requiring anti-inflammatory therapy
* Participation in previous vaccine trial
* Any component of grade 3 follicular lymphoma or transformed follicular lymphoma

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2007-06 (Actual); Primary Completion 2023-07-25 (Actual); Study Completion 2023-07-25 (Actual)

PRIMARY OUTCOMES:
To determine the safety and toxicity of administering vaccine composed of lethally irradiated lymphoma cells admixed with GM-CSF secreting K562 cells in patients with follicular lymphoma. | 2 years

SECONDARY OUTCOMES:
To describe the biologic activity of the study vaccine | 2 years
to determine tumor overall response rate as well as complete and partial response rates | 2 years
to determine progression free survival and overall survival. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Eric Jacobsen, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (1):
- Dana-Farber Cancer Institute, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Jacobsen E, Plant A, Redd R, Armand P, McDonough M, Ihuoma U, Fisher DC, LaCasce A, Ritz J, Dranoff G, Freedman A. A phase I trial of vaccination with lethally irradiated lymphoma cells admixed with granulocyte-macrophage colony-stimulating factor secreting K562 cells for the treatment of follicular lymphoma. Leuk Lymphoma. 2024 Dec;65(12):1864-1874. doi: 10.1080/10428194.2024.2381651. Epub 2024 Jul 21. PMID 39034493